CLINICAL TRIAL: NCT04747925
Title: Compare Immediate Effect Of Mulligan Two Leg Rotation And Bent Leg Raise Techniques On Hamstring Tightness And Core Muscle Weakness In Chronic Low Back Pain
Brief Title: Immediate Effect of Mulligan Two Leg Rotation and Bent Leg Raise Techniques on Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC00772 Sania Tanveer Qazi
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain; Hamstring Pulled
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan two leg rotation , core muscle strengthening exercises (Active Comparator): Group A :is receiving moist heat for the hamstrings muscles prior the Mulligan Two leg rotation technique for 10mins.Hold the position for 30 seconds, relax for 1 minute. Reps are given 3 repetitions. And 3 Sets at each session .core muscle strenthening exercises for back extensors and abdominals i.e Bridge curls ,table top ,abdominal crunches,back extension with arms supporting, is being performed. Position is being held for about 10 seconds and each exercise are performed with 10 repititions. Patient is being relaxed for 3 seconds between repetitions and 60 second rest between each exercise
  Interventions: Other: Mulligan two leg rotation core muscle strengthning exercises
- Mulligan bent leg raise technique core muscle strengthning exercises. (Experimental): Group B is receiving moist heat for the hamstrings muscles prior the Mulligan Bent leg raise technique for 10 minutes. Hold the position for 30 seconds, relax for 1 minute. Reps are 3 repetitions. And 3 Sets at each session .Subject is being receive 2 weeks protocol. core muscle strenthening exercises for back extensors and abdominals i.e Bridge curls ,table top ,abdominal crunches,back extension with arms supporting, are being performed. Position is held for about 10 seconds and each exercise is performed with 10 repititions. Patient is being relaxed for 3 seconds between repetitions and 60 second rest between each exercise
  Interventions: Other: mulligan bent leg raise technique, core muscle strengthning exercises

INTERVENTIONS:
Other: Mulligan two leg rotation core muscle strengthning exercises — Group A :is receiving moist heat for the hamstrings muscles prior the Mulligan Two leg rotation technique for 10mins.Hold the position for 30 seconds, relax for 1 minute. Reps are given 3 repetitions. And 3 Sets at each session .core muscle strenthening exercises for back extensors and abdominals i.e Bridge curls ,table top ,abdominal crunches,back extension with arms supporting, is being performed. Position is being held for about 10 seconds and each exercise are performed with 10 repititions. Patient is being relaxed for 3 seconds between repetitions and 60 second rest between each exercise
  Arms: mulligan two leg rotation , core muscle strengthening exercises
Other: mulligan bent leg raise technique, core muscle strengthning exercises — Group B is receiving moist heat for the hamstrings muscles prior the Mulligan Bent leg raise technique for 10 minutes. Hold the position for 30 seconds, relax for 1 minute. Reps are 3 repetitions. And 3 Sets at each session .Subject is being receive 2 weeks protocol. core muscle strenthening exercises for back extensors and abdominals i.e Bridge curls ,table top ,abdominal crunches,back extension with arms supporting, are being performed. Position is held for about 10 seconds and each exercise is performed with 10 repititions. Patient is being relaxed for 3 seconds between repetitions and 60 second rest between each exercise
  Arms: Mulligan bent leg raise technique core muscle strengthning exercises.

SUMMARY:
The aim of this study is to compare the immediate effect of mulligan's two leg rotation and bent leg raise for hamstring tightness, core muscle weakness in chronic low back pain, lumbar Range of motion. A randomized control trial is being conducted at Women Institute of Rehabilitation Sciences Abbottabad. It consisted of 68 participants with moderate chronic low back pain 4-6 on VAS scale, weak back extensors, and abdominal muscle weakness .and hamstring tightness. 34 patients in Group A is receiving moist heat for the hamstrings muscles prior the Mulligan Two leg rotation technique for 10mins .core muscle strenthening exercises for back extensors and abdominals. 34 patients in Group B is receiving moist heat for the hamstrings muscles prior the Mulligan Bent leg raise technique for 10 minutes.Study duration was of 6 months. Sampling technique being applied is purposive.Study includes patients with mechanical LBP more than 3 months.Tools being used in the study are Goniometer, Measuring tape, Pressure Biofeedback Unit, Visual analogue scale (VAS), Mulligan's belt. Data is being analyzed through SPSS 21.

DETAILED DESCRIPTION:
The term Low Back Pain (LBP) refers to pain in the lumbo-sacral area of the spine from 1st lumbar vertebra to the 1st sacral vertebra. Low back pain (LBP) can be caused by different varieties of problems with any parts of the complex, interconnected network of spinal muscles, nerves, bones, discs or tendons in the lumbar spine.The stability and support of the trunk area is mainly dependent on strength of supporting structures, the muscles. Weak back extensor muscles can result improper vertebral alignment which may lead to undue loading on the spine. Causes of low back pain can be due to many factors, for example: individual characteristics, working environment such as heavy physical work, awkward static and dynamic working postures, as well as manual handling and lifting, lifestyle factors and psychological factors. It can also be caused because of muscle sprain, ligament sprain, poor posture, age, disc bulge, other causes of low back pain include bladder/kidney infection, endometriosis, cancer, or ovarian problems Hamstring muscles are comprised of three semitendinosus, semimembranosus and biceps femoris. They are located on the posterior compartment of the thigh. Hamstring muscles are two joint muscles of body its function is hip extension and knee flexion. Injury rate within hamstring muscle, is the long head of biceps femoris that is frequently injured and accounts for approximately 80 % of all hamstring injuries. Flexibility is the most important component of physical fitness. Normal flexibility allows the person to move smoothly and safely . For normal movement and locomotion flexibility of muscle is important. It will help a person for normal body function. The flexibility of hamstring muscle is always emphasized more. The Hamstring muscle is the most common muscle to always go for tightness. The tightness of this muscle apparently increases from childhood up to the age of 40-49 years. Tight hamstring muscles causes a major effect on body's normal postural alignment. Till date studies have shown that tightness of hamstring always led to low back pain with lumbar intervertebral disc pathologies. Biomechanically tightness of hamstring muscle is thought to increase patellofemoral joint compressive forces because of increase in passive tension at the time of the swing phase of ambulation under rapid and stressful situations hamstring muscles fails to pass through full physiological amplitude when specifically this muscle goes for tightness.

The "core" has been described as a muscular box with the abdominals in the front, Para spinals and gluteal in the back, the diaphragm as the roof, and the pelvic floor and hip girdle musculature as the bottom. Chronic low back pain (CLBP) is a complex condition which is mainly associated with back (multifidus) abdominal (transversusabdominis) and hip (Gluteus Maximus) muscles dysfunction along with reduced lumbar flexibility Mulligan Bent Leg Raise is a newer technique which has been developed to manage hamstring tightness. This stretching technique is painless and is recently utilized in the management of hamstring tightness with limitation of straight leg raise. The Mulligan bent leg raise (BLR) technique has been described as a means of improving range of straight leg raise (SLR) in subjects with LBP and/or referred thigh pain (Mulligan, 1999). The intention of this technique is to restore normal mobility and reduce LBP and physical impairment. Impairment is defined as abnormalities of structure or function, as indicated by signs or symptoms .

Mulligan's Two Leg Rotation Technique(TLR) is also a painless technique, and it can be applied to any subjects having hamstrings tightness, low back pain or limited and/or painful straight leg raise (SLR).It can be extremely useful in patients who have a gross bilateral limitation of straight leg rising. TLR Technique is a new technique that has been developed by Dr. Brain R Mulligan and colleagues.

Toby Hall ,Sonja Hardt ,Axel Schäfer, Lena Wallin conducted a study in 2006 to investigate the immediate effects, on range of motion and pain, of Mulligan's bent leg raise (BLR) technique in subjects with limited straight leg raise (SLR) and low back pain (LBP). the study reveals that there was a significant increase in the range by 7° in the BLR group, which may be clinically important.

Pratik A. Phansopkar and Vijay Kage in 2014 conducted a study to evaluate the effectiveness of Mulligan's TLR technique for hamstrings flexibility in acute non-specific low back pain. The Results of the study were focused on Pain relief, decrease in the functional disability due to low back pain. Their study demonstrates that, Mulligan's Two Leg Rotation technique is effective in increasing the hamstrings flexibility in subjects with low back pain in terms of pain, range of motion and functional disability In 2015 Tarun Kumara, Suraj Kumarb, Md. Nezamuddinc and V.P. Sharmad conducted a study to evaluate the Efficacy of core muscle strengthening exercise in chronic low back pain patients. This study concluded that core muscle strengthening exercise is an effective rehabilitation technique for all chronic low back pain patients.

A study conducted in 2018 to investigate the Effectiveness of bent leg raise v/s two leg rotation in patients with low back pain. The study was designed to compare the immediate effects of two manual techniques in patients with low back pain. The study showed that both BLR and TLR techniques were equally effective in reducing LBP. But clinically group A bent leg raise technique showed more effective in reducing low back pain and improving ROM than group B two leg rotation.

In 2016, Parag P Kulkarni., Ankita Devasthali., Ajay Kumar and Satish Pimpale conducted a study to compare effectiveness of mulligan bent leg raise v/s knee to chest McKenzie for hamstring tightness. Their study concluded that Bend Leg raise technique of Mulligan was found to be more effective than Knee to the chest of McKenzie.

A study conducted by Shrinivas Vinayakrao Shinde, Smita Bhimrao Kanase showed that the active knee extension and straight leg raise was statistically extremely significantly improved in participants treated with mulligan bent leg raise. This improvement is mainly attributed to change in stretch tolerance of the hamstring muscle. It may also be assumed that bent leg raise triggers neurophysiological responses influencing the muscle stretch tolerance.Thus, there was improvement in active knee extension and straight leg raise range in participants.

Rina, Shamima Nasrin in 2016 conducted a study to investigate the Effectiveness of bent leg raise exercise along with conventional physiotherapy comparing with conventional physiotherapy alone for the patients with chronic radiating low back pain. Their experimental study showed that Bent Leg Raise Exercise with conventional physiotherapy was more effective than conventional physiotherapy alone for patients with chronic radiating Low Back Pain C Romani-Ruby investigated that the performance of core stability would result in increased flexibility of the hamstring musculature and vice versa. Core stability exercise programs target these muscles to help improve the overall function of the spine and body during activities of daily living, where it provides "proximal stability for distal mobility. More recent research demonstrates a significant correlation between core stability and the range of motion of the Lower extremities, specifically the hamstrings.

ELIGIBILITY:
Inclusion Criteria:

* The study includes female patients with moderate chronic low back pain 4-6 on VAS scale, weak back extensors, and abdominal muscle weakness .and hamstring tightness.
* Study included patients with mechanical LBP more than 3 months.
* Limited SLR more than 300, hamstring tightness range between 60 - 90o.

Exclusion Criteria:

* Subjects with LBP with trauma.
* LBP with specific pathology.
* Any neurological Symptoms involving prolapsed intervertebral disc, radiating pain.
* History of any recent abdominal, back Surgeries.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
ROM Hip, Knee extension | 2 weeks
  Changes from the baseline ROM of hip flexion and knee extension are being taken with the help of goniometer.
  Normal Values for Range of Motion of Hip joint in flexion with goniometer ranges from 0 -1250.
  For Active knee extension , knee flexion angle should be of greater than 150.

SECONDARY OUTCOMES:
Core muscle strength | 2 weeks and 1 month follow up
  Changes from the baseline strength of Abdominals and back extensors are being taken with the help of Pressure Biofeedback Unit. The bulb inflated to 40 mmHg of pressure and maintained .The measuring range is from 0 to 200 mmHg analog pressure with an accuracy of +/- 3mmHz pressure. pressure increase of 0, 2, 4, or 6 mmHg from the initially maintained 40 mmHg.
Visual Analogue scale | 2 weeks
  Changes from base Visual Analogue scale (VAS) is a scale for pain starting from 0-10. where 0 indicate no pain , 4 to 7 indicate mild to moderate pain and 10 indicate severe pain.
ROM lumbar spine | 2 weeks
  ROM Lumbar Spine ( Flexion) The normal ROM range for lumbar flexion ranges from 6.3cm - 6.9cm.
  ROM Lumbar Spine ( Extension ) The normal ROM range for lumbar extension ranges from 1.6cm.
  ROM Lumbar Spine ( rotation ) .normal range for rotation is 100.with measuring tape it is measured by point of marking .
  ROM Lumbar Spine ( right side bending ) The normal ROM range for lumbar SB ranges from 25 - 300.
  ROM Lumbar Spine ( left side bending) The normal ROM range for lumbar SB ranges from 25- 300.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PHD*, Principal Investigator — saira.waqar@riphah.edu.pk
Locations (1):
- Women Institute of Rehabiltation Sciences Abbottabad, Abbottabad, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinpelu AO, Bakare U, Adegoke BA. Influence of age on hamstring tightness in apparently healthy Nigerians. Journal of Nigeria Society of Physiotherapy. 2009 Jul 22; 15(2):35-41.
- [Background] Dadebo B, White J, George KP. A survey of flexibility training protocols and hamstring strains in professional football clubs in England. Br J Sports Med. 2004 Aug;38(4):388-94. doi: 10.1136/bjsm.2002.000044. PMID 15273168
- [Background] Odunaiya NA, Hamzat TK, Ajayi OF. The effects of static stretch duration on the flexibility of hamstring muscles. African journal of biomedical research. 2005;8(2):79-82.
- [Background] Nagarwal AK, Zutshi K, Ram CS, Zafar R, Hamdard J. Improvement of hamstring flexibility: A comparison between two PNF stretching techniques. International journal of sports science and engineering. 2010; 4(1):25-33.
- [Background] Phansopkar PA, Kage V. Effect of Mulligan's two leg rotation technique on hamstring flexibility in subjects with acute non-specific low back pain: clinical trial. J Med Res. 2014; 2(6):70-8.
- [Background] Kumar T, Kumar S, Nezamuddin M, Sharma VP. Efficacy of core muscle strengthening exercise in chronic low back pain patients. J Back Musculoskelet Rehabil. 2015;28(4):699-707. doi: 10.3233/BMR-140572. PMID 25467999
- [Background] Shinde SV, Kanase SB. Effect of Mulligan Bent Leg Raise versus Neural Mobilization on Hamstring Tightness in College Students. Iosr Journal of Dental and Medical Sciences. 2017 Mar; 16:3-59.